CLINICAL TRIAL: NCT02250989
Title: Influence of Glycaemia and Insulinemia on Vasomotor Endothelial Function After Ischemia/Reperfusion Lesion on Patients in Acute Phase of ST Segment Elevation Myocardial Infarction (STEMI)
Brief Title: The Influence of Glycaemia and Insulinemia on Vasomotor Endothelial Function After Myocardial Infarction
Acronym: INGLIVEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Assistent Professor, Cardiology Division, University of Campinas, Brazil
Other Study IDs: Ateroloab-1
Record Dates: First submitted 2014-09-22; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Myocardial Infarction
Keywords: Endothelial disfunction; Intercellular Adhesion Molecule-1; Vascular Cell Adhesion Molecule-1; 8-epi-prostaglandin F2alpha; Nitric Oxide; Plasminogen Activator Inhibitor 1; Endothelin-1; Tumor Necrosis Factor-alpha; Glucose; Insulin; C-peptide; C-reactive protein; 3-nitrotyrosine
MeSH Terms: conditions — Myocardial Infarction; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, whole blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hyperinsulinemia/Euglycaemia: In this group study, a condition of Hyperinsulinemia/Euglycaemia will be held trough clamp study, during witch FMD will be measured before and after ischemia/reperfusion injury.
- Hyperinsulinemia/Hyperglycemia: In this group study, a condition of Hyperinsulinemia/Hyperglycemia will be held trough clamp study, during witch FMD will be measured before and after ischemia/reperfusion injury.
- Hypoinsulinemia/Hyperglycemia group: In this group study, a condition of Hypoinsulinemia/Hyperglycemia will be held trough clamp study, during witch FMD will be measured before and after ischemia/reperfusion injury.

SUMMARY:
The objective of this study is to investigative the influence of different levels of glycaemia or insulinemia in vascular endothelium in ischemia/reperfusion lesion after myocardial infarction

DETAILED DESCRIPTION:
The study will include patients consecutively admitted with acute myocardial infarction at State University of Campinas Hospital. Participants will be evaluated during hospitalization and, after they fulfill the inclusion criteria and sign an informed consent, it will be collected a brief medical history and recorded results from glycated hemoglobin (HbA1c), glycaemia, total cholesterol (TC), triglycerides (TG), HDL cholesterol (HDL-C), C-reactive protein (CRP), urea (U), creatinine (Cr), markers of myocardial necrosis (troponin T and CK-MB), Hemoglobin, Red blood cell, Leucocytes, Na, K, Ca and Mg.

In the first week after infarction, from admission until the realization of the clamps experiments (the medical procedure where blood glucose and insulin levels will be controlled), all medications prescribed, medical history and examination will be recorded, as well as follow-up during hospitalization.

At the day of the clamp, between 144 and 168 hours after infarction, volunteers will be randomized to one of the three situations with different glycemic and insulinemic conditions, i.e., a) high insulinemia and low glycaemia, b) high insulinemia and high glycaemia and c) low insulinemia and high glycaemia. During these experiments, endothelial vasomotor function will be recorded in four periods: i) before initiation of the procedure, ii) after 1h of the beginning, iii) 30 minutes after the second procedure and iv) 15 minutes after the simulation of ischemia/reperfusion lesion. In each time point, the investigators will collect plasma to dose inflammatory, oxidative stress and vascular activation markers.

Hospital care of subjects

The patients included in this survey will be treated according to actual guidelines. Briefly, will be enrolled patients who underwent primary angioplasty within 6 hours after symptoms onset, were introduced antiplatelet and anticoagulation therapy at the correct dose, respectively Acetylsalicylic Acid (ASA) 200 mg and Clopidogrel 300 mg, and enoxaparin 30 mg. In patients without contraindication, it will be administered in the first 24 hours beta-blockers and ACEi in those with ejection fraction (EF) <0.4, previous MI or prior heart failure. Upon admission, if there is no contraindication, simvastatin 40 mg/day will be administered. As a maintenance dose, the investigators will administer ASA 100 mg, clopidogrel 75 mg, enoxaparin 1 mg/kg twice daily, simvastatin 40 mg, propranolol 40 mg or metoprolol 50 mg (beta-blockers available at the hospital) and captopril 25 mg (most used ACEi). Patients will be treated preferably in the Coronary Unit (CU). Researchers may suggest the physician responsible for the patient care to prescribe the above medications, as well as question why the drugs listed in the guidelines are not being used. The reasons and specific contraindications will be recorded.

The researchers are not directly responsible for the treatment of individuals, which does not absolve them of responsibility for any adverse effects related to the experiments. Also, the investigators emphasize that the study did not interfere with the flow of patients during hospitalization, i.e., will not influence the discharge of patients.

Randomization to one of the three clamps

As observed, the investigators will evaluate endothelial reactivity by FMD. On the day of the clamp, after fasting, they will be exposed to one of three situations: (i) hyperglycemia / hypoinsulinemia, (ii) euglycaemia / hyperinsulinemia and (iii) hyperglycemia / hyperinsulinemia.

The clamps will simulate the possible attenuation or increase in endothelial reactivity promoted by the independent variables during ischemia/reperfusion (I/R) injury. In total, the test will consist of realization of a basal FMD-1 (during 15 minutes), clamps (variable length, usually 60 minutes), FMD-2 (15 min) after the clamp, rest time (30 min), ischemia/reperfusion (20 min) injury, rest time (15 min) and FMD-3 (15 min). Throughout the experiment, blood glucose and insulin will be controlled and maintained at levels such as designed previously for each clamp situation. In all subjects, plasma samples will be collected before the start of the clamp (during FMD-1), at the end of the measurement of the second FMD during the clamp, prior to the I/R injury and 15 minutes after the end of the same test (during FMD-3). In these samples will be dosed insulin, glucose, C-peptide, C-reactive protein, tumor necrosis factor-α (TNF-α), nitric oxide, intercellular adhesion molecule-1 (ICAM-1), plasminogen activator inhibition-1 (PAI-1), isoprostane and interleucin-1 (IL-1).

In one group, the euglycemic/hyperinsulinemic consists of a situation in which insulin levels are above physiological levels and blood glucose levels maintained at approximately 100 mg/dL. Euglycemic/hyperinsulinemic clamp is similar to the way the hyperinsulinemic/hyperglycemic clamp is performed, although reaching a glucose level of approximately 150 mg/dL. During the clamp with hypoinsulinemia/hyperglycemia, will be infused a somatostatin analogue (octreotide) for 30 minutes (t = 0 min) and subsequently infusion of 20% glucose to achieve glycaemia of approximately 150 mg/dL (t = 30 min).

Ischemia/Reperfusion Injury The I/R injury is intended to simulate at the brachial artery a condition similar to coronary lesion resulting from infarction after reperfusion. This experiment will be performed 30 min after the measurement of FMD-2, positioning a pneumatic cuff at level of brachial artery, inflating it to 200 mmHg for 15 minutes. After this period of ischemia, the cuff is deflated and is subsequently performed the brachial reactivity test. This ischemia period is safe, as shown in other studies.

Statistical analysis Data will presented as mean ± standard deviation (SD) when normally distributed or median and interquartile range (IQR) for non-normal data. Categorical variables will be compared by chi-square. Continuous variables with normal distribution will be compared using analysis of covariance (ANCOVA) adjusted for age, gender, size of MI estimated by peak CK-MB and estimated by heart rate variability sympathetic activity. Prerequisites for the ANCOVA models (linearity, normality and equal variance) will be checked using histograms, normal probability plots and residual dispersion. Non-normal continuous variables may be transformed logarithmically. If, after the transformation, they persist not normal, will be analyzed by the Kruskal-Wallis test. Analysis will be performed using the SPSS 22 application, Mac version.

ELIGIBILITY:
Inclusion Criteria:

* less than 12 hours from the onset of symptoms of STEMI,
* reperfusion therapy performed less than 6 hours of symptom onset.

Exclusion Criteria:

* patients that after 24 hours did not show markers of myocardial necrosis
* diabetes or use of oral antidiabetics
* admission with glycosylated hemoglobin ≥ 6.5%
* patients with creatinine clearance <50 ml / min,
* patients with BMI ≥ 40 kg / m2,
* premenopausal women,
* patients that used nitrate or vasoactive drugs (norepinephrine, dobutamine, nitroglycerin or nitroprussiate in 48h prior to the examination of endothelial function
* cardiac dysfunction in acute MI with or without repercussion clinic, diagnosed by ejection fraction less than 50% left ventricle.
* FMD values above or below 2 standard deviations or more from the average of these tests

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with ST segment elevation myocardial infarction (STEMI) attended at Clinics Hospital of Campinas
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change in endothelial function after ischemia/reperfusion injury | Between 144 and 168 h after Myocardial Infarction
  Compare the effects of euglycemic/hyperinsulinemic, hyperglycemic/hypoinsulinemic and hyperglycemic/hyperinsulinemic on endothelial reactivity, measured by flow mediated dilation, after ischemia/reperfusion injury assessed at brachial artery.

SECONDARY OUTCOMES:
Change in plasma pool of nitric oxide after ischemia/reperfusion injury | Between 144 and 168 h after Myocardial Infarction
  Compare the effects of euglycemic/hyperinsulinemic, hyperglycemic/hypoinsulinemic and hyperglycemic/hyperinsulinemic on nitric oxide generation before and after ischemia/reperfusion injury assessed at brachial artery.
Change in inflammatory markers after ischemia/reperfusion injury | Between 144 and 168 h after Myocardial Infarction
  Compare the effects of euglycemic/hyperinsulinemic, hyperglycemic/hypoinsulinemic and hyperglycemic/hyperinsulinemic on markers of inflammatory activity (CRP, TNF alpha, IL-1 beta and IL-10) in after ischemia/reperfusion injury assessed at brachial artery.
Change in biomarkers of endothelial dysfunction before and after ischemia/reperfusion injury | Between 144 and 168 h after MI
  Compare the effects of euglycemic/hyperinsulinemic, hyperglycemic/hypoinsulinemic and hyperglycemic/hyperinsulinemic on markers of endothelial activation (ICAM-1, VCAM-1, PAI-1) in after ischemia/reperfusion injury assessed at brachial artery.
Change in biomarkers of oxidative stress before and after ischemia/reperfusion injury | Between 144 and 168h after MI
  Compare the effects of euglycemic/hyperinsulinemic, hyperglycemic/hypoinsulinemic and hyperglycemic/hyperinsulinemic on markers of oxidative stress (nitrotyrosine and 8-isoprostane) before and after ischemia/reperfusion injury assessed at brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, PhD, MD, Principal Investigator — Cardiology Division, Campinas State University
Locations (1):
- Clinics Hospital, Campinas, São Paulo, Brazil